CLINICAL TRIAL: NCT01027767
Title: Effect of Surgery and Radiation Therapy on Tc-99M Sestamibi Uptake Patterns in Molecular Breast Imaging
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Nicole P. Sandhu, MD, PhD, Mayo Clinic
Other Study IDs: 09-000455
Record Dates: First submitted 2009-12-08; First posted 2009-12-09 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2012-02

CONDITIONS: Breast Cancer
Keywords: Breast; MBI; Molecular; Molecular Breast Imaging; Dense breast tissue; Surgery; Radiation; BCT
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Surgery/Radiation Arm: Patients that have had surgery along with radiation therapy
  Interventions: Device: Molecular Breast Imaging
- Surgery Arm: Patients that have had surgery of a benign lesion.
  Interventions: Device: Molecular Breast Imaging

INTERVENTIONS:
Device: Molecular Breast Imaging — Molecular Breast Imaging

SUMMARY:
The investigators hope to prove that radiation and surgical scarring does not result in changes that affect the MBI pattern 6-12 months after completion of treatment.

DETAILED DESCRIPTION:
The study will allow us to evaluate whether surgery and radiation have persistent effects on the breast tissue with regards to whether and how such changes impact MBI images and to determine whether the inflammatory changes due to treatment resolve within 6-12 months of completing treatment.

ELIGIBILITY:
Inclusion Criteria:

* Women who have planned surgical excision of a lesion or have had a baseline MBI study as part of another MBI research protocol who are within 6-12 months of completing breast surgery who are able and willing to return to Mayo Clinic for a follow up MBI study once the 6-12 month interval is complete.
* Women who plan BCT for a malignant lesion or who are within 6-12 months of completing breast conserving treatment and have had a baseline MBI study as part of another MBI research protocol and are able and willing to return to Mayo Clinic for a follow up MBI study.

Exclusion Criteria:

* Women who do not require surgical excision of a breast lesion or breast conserving treatment for breast cancer.
* Patients undergoing mastectomy.
* Women who are pregnant or lactating.
* Women who are taking hormonal contraception or hormone replacement therapy (vaginal estrogen is permitted), or have used these agents within the previous 3 months.
* Women who have received chemotherapy within the previous 6 months or receive chemotherapy as part of their cancer treatment.
* Men (due to the very low incidence of male breast cancer and the lack of any available data regarding the use of scintimammography or MBI in men).
* Women under the age of 18 years.
* Women unable to sit comfortably during image acquisition.
* Women who are unable to return to Mayo Clinic for a follow up MBI scan 6-12 months after surgical excision or 6-12 months after completing radiation therapy for breast conservation.

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women who are seen in the Mayo Clinic Breast Clinic
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2009-05; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Sandhu, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States